CLINICAL TRIAL: NCT04618588
Title: Evaluation of Computer-guided Low Window Sinus Lift Technique (A Clinical Trial)
Brief Title: Computer Guided Low Window Sinus Lift Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sinus lift
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Sinus Perforation
Keywords: sinus augmentation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sinus elevation using "Low Window Sinus Lift" technique (Experimental)
  Interventions: Procedure: Low Window Sinus Lift technique

INTERVENTIONS:
Procedure: Low Window Sinus Lift technique — Preoperative CBCT of surgical site and Fabrication CAD/CAM surgical stent, Sinus elevation using "Low Window Sinus Lift" technique, Implant, bone graft and membrane placement

SUMMARY:
The study group included 12 patients that were treated using the low window lateral sinus lift technique with simultaneous implant placement. This was facilitated using a CAD-CAM generated surgical guide. Subjective assessment on postoperative pain and swelling as well as objective assessment of implant stability, vertical bone height gained and complications such as Schneiderian membrane perforation rates and bleeding.

DETAILED DESCRIPTION:
Presurgical assessment of each patient was performed. Preoperative impressions were taken and study models were mounted. Orthopantogram (OPG) and cone beam computer tomography (CBCT) of the targeted areas were also done in order to evaluate residual bone height between the alveolar bone crest and the sinus floor, residual ridge width, bone quality and planning the number, size and position the implants.

Designing the surgical guide was performed using In2Guide™ system powered by OnDemand3D™.

The low window design was also planned where the lower osteotomy line will be flushed with the floor of the sinus, the upper line is 6mm of height from the lower line, the mesial line is flushed with the anterior wall and the distal line will correspond to the position of the most distal implant. The final product was fabricated using OnDemand3D™ which was then transferred to the 3d printer machine.

Patients were instructed to rinse with 0.125% chlorhexidine antiseptic mouth-wash for 2 minutes prior to surgery. The surgical area was anesthetized with local anesthesia. Infraorbital and greater palatine nerve blocks and local infiltration were given in order to properly anesthetize the area. A crestal incision was made in the posterior edentulous area followed by a vertical incision made at 45 degrees distal to the most anterior tooth. A full thickness mucoperiosteal flap was elevated at the surgical site enabling the apical osteotomy line to be drawn at a distance of 6mm above the residual bone height from the ridge. The customized surgical guide was secured in its proper position. After drilling, the anchor pin was placed in the prepared place. Using the standardized piezoelectric tip (SL1) with sterile saline irrigation, the outline of the window in the lateral maxillary sinus wall was formed.

The bone window was thinned down using the specialized DASK drill #4 and #5 from the DASK Kit until the grey shadow of the sinus membrane becomes visible. The sinus membrane at the circumference of the bony window was detached using the dome-shaped Sinus Membrane Elevator (XSE1L). Sinus membrane elevators (XSE2L), (XSE3L) and (XSE4L) were used to carefully lift the sinus membrane from the floor and anterior wall of the sinus to create adequate space for graft material (Figure 2-b). The membrane was further elevated to the medial wall in order to provide additional blood supply from that bone. The implants were drilled in the positions indicated by the surgical guide. Half the amount of the xenograft was introduced into the cavity followed by insertion of the dental implants. The dental implants were placed at torque 30~45N‧cm. Stability of the implants was measured using an implant stability meter.

Filling the cavity with the rest of the xenograft was completed after implant placement(s). The size of the collagen membrane was adjusted to match the size of the lateral bone window and then placed and stabilized by the cover screw. The flap was released by short horizontal cuts in the inner surface of the mucosa to provide a tension free flap. This was followed by closure of the flap with water tight sutures (horizontal mattress with a single interrupted it's centre) using 3/0 silk suture material.

After 6 months from the operation, a small incision was made directly over the implant and the cover screw was removed. Implant stability was measured again using the Osstell device. The abutment was placed at torque 25~30 N.cm. An impression was taken and sent to the lab for fixed prosthetics construction. The fixed prosthesis was cemented using glass ionomer cement.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring implant placement in the posterior maxilla (Kennedy Classification: Class 1 and Class 2).
* Age between 20-60 years irrespective of the gender.
* Tooth extractions at the implant sites were performed at least 4 months before surgery.
* Residual bone height between the alveolar bone crest and the sinus floor ranges from 4 to 6 mm.
* Patients who are willing and fully capable to comply with the study protocol.

Exclusion Criteria:

* Maxillary sinus pathologies (sinusitis, long standing nasal obstruction).
* Any disease contraindicating surgery (e.g. uncontrolled diabetes).
* Heavy smokers.
* Acute oral infections.
* Untreated periodontal disease.
* Poor oral hygiene.
* A history of radiotherapy or chemotherapy of the head and neck region.
* Pregnancy.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Presence or absence of intra or postoperative complications | 6 months
  * Schneiderian membrane perforation occurrence is noted intraoperatively
  * Intra/post operative bleeding, postoperative sinusitis, periimplantitis
Postoperative pain | 1 week
  This was assessed using a 10-point Visual Analogue Scale (VAS) in the 1st week postoperatively.
  (0-1=None, 2-4=Mild-Moderate, 8-10= Severe)

SECONDARY OUTCOMES:
Implant stability | 6 months
  Implant stability is measured using the Osstell device immediately following implant placement and 6 months postoperatively (prior to abutment loading).
Postoperative edema | 1 week
  This was assessed in the 1st week postoperatively and measured as follows:
  * None (no inflammation)
  * Mild (intraoral swelling confined to the surgical field)
  * Moderate (extraoral swelling in the surgical zone)
  * Severe (extraoral swelling spreading beyond the surgical zone)+
Bone Density | 6 months
  Radiographic evaluation of bone density around each implant was done using OnDemand3D™ program.
  Measurements were taken as follows:
  1. From the tool bar, the bone density around the implant was selected from task section.
  2. The required area was selected and bone density was chosen. Mean, standard deviation, minimum and maximum readings were automatically displayed by the system.
Vertical bone height gained | 6 months
  4 reference points are selected on the CBCT. A vertical line immediately adjacent to the implant threads perpendicular to the horizontal line is drawn to a point on the bony floor of the maxillary sinus. From the cross-sectional view of 6 months postoperative, the distance from the crestal bone at the implant platform and the bone apical to the implant apex. The measurements are then subtracted from the preoperative bone height to obtain the amount of vertical bone height gained.
Marginal bone loss | 6 months
  Marginal bone loss (MBL) were measured at the buccal and palatal aspects of each implant using the implant/abutment junction as a reference point to the most coronal bone-implant junction. Measurements were performed on the CBCT immediately after surgery (baseline) and 6 months postoperatively.
  A decrease in this vertical distance between the reference point and the most coronal bone-implant contact on consecutive radiographs indicated a marginal bone loss (MBL).

CONTACTS AND LOCATIONS:
Overall Officials: Nagy H Elprince, pHd, Study Director — Alexandria University; Riham M Fliefel, pHd, Study Director — Alexandria University
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aghaloo TL, Misch C, Lin GH, Iacono VJ, Wang HL. Bone Augmentation of the Edentulous Maxilla for Implant Placement: A Systematic Review. Int J Oral Maxillofac Implants. 2016;31 Suppl:s19-30. doi: 10.11607/jomi.16suppl.g1. PMID 27228250
- [Background] Antonaya-Mira R, Barona-Dorado C, Martinez-Rodriguez N, Caceres-Madrono E, Martinez-Gonzalez JM. Meta-analysis of the increase in height in maxillary sinus elevations with osteotome. Med Oral Patol Oral Cir Bucal. 2012 Jan 1;17(1):e146-52. doi: 10.4317/medoral.16921. PMID 22157659
- [Background] Antonoglou GN, Stavropoulos A, Samara MD, Ioannidis A, Benic GI, Papageorgiou SN, Sandor GK. Clinical Performance of Dental Implants Following Sinus Floor Augmentation: A Systematic Review and Meta-Analysis of Clinical Trials with at Least 3 Years of Follow-up. Int J Oral Maxillofac Implants. 2018 May/Jun;33(3):e45-e65. doi: 10.11607/jomi.6417. PMID 29763503
- [Background] Bornstein MM, Cionca N, Mombelli A. Systemic conditions and treatments as risks for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:12-27. PMID 19885432
- [Background] Boyne PJ, James RA. Grafting of the maxillary sinus floor with autogenous marrow and bone. J Oral Surg. 1980 Aug;38(8):613-6. No abstract available. PMID 6993637
- [Background] Cavalcanti MC, Guirado TE, Sapata VM, Costa C, Pannuti CM, Jung RE, Cesar Neto JB. Maxillary sinus floor pneumatization and alveolar ridge resorption after tooth loss: a cross-sectional study. Braz Oral Res. 2018 Aug 6;32:e64. doi: 10.1590/1807-3107BOR-2018.vol32.0064. PMID 30088551
- [Background] Cosci F, Luccioli M. A new sinus lift technique in conjunction with placement of 265 implants: a 6-year retrospective study. Implant Dent. 2000;9(4):363-8. doi: 10.1097/00008505-200009040-00014. PMID 11307560
- [Background] Danesh-Sani SA, Loomer PM, Wallace SS. A comprehensive clinical review of maxillary sinus floor elevation: anatomy, techniques, biomaterials and complications. Br J Oral Maxillofac Surg. 2016 Sep;54(7):724-30. doi: 10.1016/j.bjoms.2016.05.008. Epub 2016 May 25. PMID 27235382
- [Background] Dula K, Mini R, van der Stelt PF, Buser D. The radiographic assessment of implant patients: decision-making criteria. Int J Oral Maxillofac Implants. 2001 Jan-Feb;16(1):80-9. PMID 11280366
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fugazzotto PA. The modified trephine/osteotome sinus augmentation technique: technical considerations and discussion of indications. Implant Dent. 2001;10(4):259-64. doi: 10.1097/00008505-200110000-00009. PMID 11813667
- [Background] Hwang D, Wang HL. Medical contraindications to implant therapy: Part II: Relative contraindications. Implant Dent. 2007 Mar;16(1):13-23. doi: 10.1097/ID.0b013e31803276c8. PMID 17356368
- [Background] Jivraj S, Chee W. Treatment planning of implants in posterior quadrants. Br Dent J. 2006 Jul 8;201(1):13-23. doi: 10.1038/sj.bdj.4813766. PMID 16829878
- [Background] Johnson C. Measuring Pain. Visual Analog Scale Versus Numeric Pain Scale: What is the Difference? J Chiropr Med. 2005 Winter;4(1):43-4. doi: 10.1016/S0899-3467(07)60112-8. PMID 19674646
- [Background] Liddelow G, Klineberg I. Patient-related risk factors for implant therapy. A critique of pertinent literature. Aust Dent J. 2011 Dec;56(4):417-26; quiz 441. doi: 10.1111/j.1834-7819.2011.01367.x. PMID 22126353
- [Background] Lum AG, Ogata Y, Pagni SE, Hur Y. Association Between Sinus Membrane Thickness and Membrane Perforation in Lateral Window Sinus Augmentation: A Retrospective Study. J Periodontol. 2017 Jun;88(6):543-549. doi: 10.1902/jop.2017.160694. Epub 2017 Feb 26. PMID 28398119
- [Background] Mandelaris GA, Rosenfeld AL. A novel approach to the antral sinus bone graft technique: the use of a prototype cutting guide for precise outlining of the lateral wall. A case report. Int J Periodontics Restorative Dent. 2008 Dec;28(6):569-75. PMID 19146052
- [Background] Marin S, Kirnbauer B, Rugani P, Payer M, Jakse N. Potential risk factors for maxillary sinus membrane perforation and treatment outcome analysis. Clin Implant Dent Relat Res. 2019 Feb;21(1):66-72. doi: 10.1111/cid.12699. Epub 2018 Nov 26. PMID 30475442
- [Background] Monje A, Monje F, Gonzalez-Garcia R, Suarez F, Galindo-Moreno P, Garcia-Nogales A, Wang HL. Influence of atrophic posterior maxilla ridge height on bone density and microarchitecture. Clin Implant Dent Relat Res. 2015 Feb;17(1):111-9. doi: 10.1111/cid.12075. Epub 2013 Apr 22. PMID 23607367
- [Background] Osman AH, Mansour H, Atef M, Hakam M. Computer guided sinus floor elevation through lateral window approach with simultaneous implant placement. Clin Implant Dent Relat Res. 2018 Apr;20(2):137-143. doi: 10.1111/cid.12559. Epub 2017 Dec 1. PMID 29194927
- [Background] Pal US, Sharma NK, Singh RK, Mahammad S, Mehrotra D, Singh N, Mandhyan D. Direct vs. indirect sinus lift procedure: A comparison. Natl J Maxillofac Surg. 2012 Jan;3(1):31-7. doi: 10.4103/0975-5950.102148. PMID 23251055
- [Background] Sennerby L, Meredith N. Implant stability measurements using resonance frequency analysis: biological and biomechanical aspects and clinical implications. Periodontol 2000. 2008;47:51-66. doi: 10.1111/j.1600-0757.2008.00267.x. No abstract available. PMID 18412573
- [Background] Shah SA, Khan I, Shah HS. Effectiveness of submucosal dexamethasone to control postoperative pain & swelling in apicectomy of maxillary anterior teeth. Int J Health Sci (Qassim). 2011 Jul;5(2):156-65. PMID 23267293
- [Background] Simsek Kaya G, Daltaban O, Kaya M, Kocabalkan B, Sindel A, Akdag M. The potential clinical relevance of anatomical structures and variations of the maxillary sinus for planned sinus floor elevation procedures: A retrospective cone beam computed tomography study. Clin Implant Dent Relat Res. 2019 Feb;21(1):114-121. doi: 10.1111/cid.12703. Epub 2018 Dec 17. PMID 30556642
- [Background] Stacchi C, Andolsek F, Berton F, Perinetti G, Navarra CO, Di Lenarda R. Intraoperative Complications During Sinus Floor Elevation with Lateral Approach: A Systematic Review. Int J Oral Maxillofac Implants. 2017 May/Jun;32(3):e107-e118. doi: 10.11607/jomi.4884. PMID 28494033
- [Background] Stern A, Green J. Sinus lift procedures: an overview of current techniques. Dent Clin North Am. 2012 Jan;56(1):219-33, x. doi: 10.1016/j.cden.2011.09.003. PMID 22117952
- [Background] Summers RB. A new concept in maxillary implant surgery: the osteotome technique. Compendium. 1994 Feb;15(2):152, 154-6, 158 passim; quiz 162. PMID 8055503
- [Background] Sverzut AT, Stabile GA, de Moraes M, Mazzonetto R, Moreira RW. The influence of tobacco on early dental implant failure. J Oral Maxillofac Surg. 2008 May;66(5):1004-9. doi: 10.1016/j.joms.2008.01.032. PMID 18423293
- [Background] Tatum H Jr. Maxillary and sinus implant reconstructions. Dent Clin North Am. 1986 Apr;30(2):207-29. PMID 3516738
- [Background] Tatum OH Jr, Lebowitz MS, Tatum CA, Borgner RA. Sinus augmentation. Rationale, development, long-term results. N Y State Dent J. 1993 May;59(5):43-8. PMID 8510868
- [Background] Trombelli L, Franceschetti G, Rizzi A, Minenna P, Minenna L, Farina R. Minimally invasive transcrestal sinus floor elevation with graft biomaterials. A randomized clinical trial. Clin Oral Implants Res. 2012 Apr;23(4):424-32. doi: 10.1111/j.1600-0501.2011.02318.x. Epub 2011 Oct 21. PMID 22092804
- [Background] Wilson TG Jr, Nunn M. The relationship between the interleukin-1 periodontal genotype and implant loss. Initial data. J Periodontol. 1999 Jul;70(7):724-9. doi: 10.1902/jop.1999.70.7.724. PMID 10440632
- [Background] Zaniol T, Zaniol A. A Rational Approach to Sinus Augmentation: The Low Window Sinus Lift. Case Rep Dent. 2017;2017:7610607. doi: 10.1155/2017/7610607. Epub 2017 Feb 26. PMID 28337349
- [Background] Zaniol T, Zaniol A, Tedesco A, Ravazzolo S. The Low Window Sinus Lift: A CAD-CAM-Guided Surgical Technique for Lateral Sinus Augmentation: A Retrospective Case Series. Implant Dent. 2018 Aug;27(4):512-520. doi: 10.1097/ID.0000000000000776. PMID 29847458
- [Background] Zitzmann NU, Margolin MD, Filippi A, Weiger R, Krastl G. Patient assessment and diagnosis in implant treatment. Aust Dent J. 2008 Jun;53 Suppl 1:S3-10. doi: 10.1111/j.1834-7819.2008.00036.x. PMID 18498582